CLINICAL TRIAL: NCT04231357
Title: Great Trochanteric Pain Syndrome: Parallel Group, Blind Randomised Clinical Trial to Assess the Efficacy and Safety of PRP Injection Versus Needle Tenotomy With Lidocaine
Brief Title: Greater Trochanteric Pain Syndrome: Efficacy of Ultrasound Guided Platelet-rich Plasma vs Needle Tenotomy.
Acronym: PRP-GTPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isabel Andia (Other Government)
Responsible Party: Sponsor-Investigator, Isabel Andia, Ph.D., Basque Health Service
Organization: Basque Health Service (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-GTPS; 2019-000538-21 (EudraCT Number)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Tendinopathy
Keywords: ultrasound;platelet-rich plasma;tendinopathy;pain;trochanter
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: Single center, superiority type, double blinded, randomised controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: blocks of four, using EPIDAT3.1 statistical program, and created aluminum paper blinded envelopes with the numbered treatment allocation. The numbered envelopes will be opened on the treatment day by the researcher who is in charge of the PRP preparation. All physicians (including orthopaedists involved in clinical outcome assessments and radiologists involved in ultrasound assessments), except one radiologist who performed the procedures, will be unaware of treatment allocation. All patients will be blinded to the treatment. Peripheral blood will be drawn from all patients, and the syringe containing the treatment will be wrapped with gauze hindering treatment visualization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma (PRP) (Experimental): 3 mL of autologous platelet rich plasma with a moderate concentration of platelet (2x above peripheral blood) and no leukocytes will be injected under ultrasound guidance
  Interventions: Drug: platelet rich plasma
- control (Active Comparator): needle tenotomy with lidocaine
  Interventions: Drug: platelet rich plasma

INTERVENTIONS:
Drug: platelet rich plasma — platelet rich plasma prepared from peripheral blood using single spin centrifugation
  Other Names: PRP

SUMMARY:
Great trochanteric pain syndrome (GTPS) is a difficult problem to manage and results in significant patient morbidity. This study is a single-center, randomized double-blind controlled trial. Eighty patients will be allocated to have an ultrasound (US)-guided injection of pure platelet-rich plasma (PRP) or needle tenotomy. Outcome data will be collected before the intervention, and at 3, 6, and 12 months after intervention. Main outcome measure: percent of patients that experience a reduction of 25% in hip outcome score (HOS) (responders) at 6 months after the intervention. Secondary outcome measures include percent of responders at three and twelve months, and pain reduction (VAS) at 3, 6, and 12 months. Adverse reactions or events will be recorded.

DETAILED DESCRIPTION:
Evaluation of gluteal tendon pathology, including superoposterior and lateral aspects of gluteus medius and gluteus minimus(changes in echotexture, partial tears, calcified deposits, thickness, and loss of fibrillar pattern were evaluated by ultrasound at baseline, six and 12 m post-treatment. Peritrochanteric pathology including tensor fascia lata, trochanteric bursa, and cortical irregularities were also recorded. To analyze the relationship between the possible predictor variables (including sociodemographic and clinical factors, and imaging biomarkers, such as tendon degeneration and abnormalities in the peritrochanteric space) and changes in pain (VAS score) and functionality (HOS score), multivariate analyses were performed using multiple linear regressions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between the ages of 35 and 75 years.
* At the screening visit, they present hip pain at 3 points out of 10 in EVA.
* Body Mass Index values between 20 and 35 (both values included).
* Commitment to comply with all study procedures.
* Diagnoses of chronic GTPS according to the diagnostic criteria that have been previously described.
* The patient must give written informed consent.
* Women of child-bearing age must obtain a negative test result of pregnancy in blood or urine and accept the use of appropriate contraception while in the trial.

Exclusion Criteria:

* • Body Mass Index>35.

  * Presence of full tendon tear.
  * Systemic autoimmune rheumatologic disease (connective tissue diseases and systemic necrotizing vasculitis)
  * Poorly controlled diabetes mellitus (glycosylated hemoglobin above 9%)
  * Blood disorders (thrombopathy, thrombocytopenia, anemia with Hb <9)
  * Patients receiving immunosuppressive treatments
  * Treatment by intramuscular corticoid, during the 3 months prior to the first administration of the trial treatment.
  * Treatment with non-steroidal anti-inflammatory drugs (more than 10 days consecutive to usual doses), opiates or oral steroids during the 15 days prior to treatment in the study.
  * Severe heart disease
  * Patients unable to comply with scheduled visits, for work or spend long periods away from their habitual residence.
  * Patients with active cancer or cancer diagnosed in the last five years.
  * Analytical Diagnosis Hepatitis B, C or HIV infection.
  * Pregnant or lactating.
  * People who are taking a drug in clinical investigation or participated in any investigational study clinic (with an authorized or not) within 30 days prior to randomization.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Rate of participants that showed a clinically minimal clinically important change in function as measured by HOS (Hip Outcome Score, Activity of Daily Living Scale) | 6 months
  Rate of participants that experience at least 25% change in Hip Outcome score (HOS) (comparing to baseline) (Hip Outcome Score, Activity of Daily Living Scale, 0 (worst) to 100 (level of activity prior to hip problem)
Number of adverse events related to treatment | 3 months
  Differences in the patient self-reported adverse events related to treatment

SECONDARY OUTCOMES:
Rate of patients that experience a significant minimal clinically important change in HOS at 3 and 12 months | 3 and 12 months
  Rate of patients that experience at least 25% change in Hip Outcome score (HOS, Activity of Daily Living Scale, 0 to 100 (level of activity prior to hip problem)
Pain changes (VAS) (0 to 10 maximum pain) | 3, 6 and 12 months
  Pain changes assessed by visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Cruces University Hospital, Barakaldo, Bizkaia, Spain

REFERENCES:
- [Result] Atilano L, Martin N, Ignacio Martin J, Iglesias G, Mendiola J, Bully P, Aiyegbusi A, Manuel Rodriguez-Palomo J, Andia I. Ultrasound-Guided Subfascial Platelet-Rich Plasma Injections Versus Enthesis Needling for Greater Trochanteric Pain Syndrome: A Randomized Controlled Trial. Orthop J Sports Med. 2024 May 14;12(5):23259671241249123. doi: 10.1177/23259671241249123. eCollection 2024 May. PMID 38751852
- See also: here is a link to the open access article containing the clinical trial results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC11095191/